CLINICAL TRIAL: NCT01946568
Title: A Phase 1, Open Label, Single Dose Study To Investigate The Pharmacokinetics, Safety and Tolerability Of Dalbavancin In Hospitalized Children Aged 3 Months to 11 Years Receiving Standard Intravenous Anti-Infective Treatment For Bacterial Infections
Brief Title: A Single Dose Study To Investigate The Pharmacokinetics and Safety Of Dalbavancin In Hospitalized Children Aged 3 Months to 11 Years.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Durata Therapeutics Inc., an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DUR001-106
Record Dates: First submitted 2013-08-29; First posted 2013-09-19 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Bacterial Infections.
MeSH Terms: conditions — Bacterial Infections | interventions — dalbavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single dose Dalbavancin (Experimental)
  Interventions: Drug: Dalbavancin

INTERVENTIONS:
Drug: Dalbavancin — Intravenous dalbavancin given at 15 mg/kg (not to exceed 1000 mg) for patients ≥5 years of age, and 25 mg/kg for patients <5 years of age.

SUMMARY:
A phase one study to characterize the pharmacokinetics of dalbavancin in pediatric patients aged 3 months to 11 years (inclusive) following the intravenous administration of a single dose of dalbavancin.

DETAILED DESCRIPTION:
This is a open label, multi center study to investigate the pharmacokinetics, safety and tolerability of a single dose of intravenous dalbavancin in hospitalized pediatric patients with known or suspected bacterial infection. Patients will be enrolled and results will be evaluated in 3 age cohorts as follows:

Cohort 1: Patients 6 years to 11 years of age, inclusive; Cohort 2: Patients 2 years to <6 years of age; Cohort 3: Patients 3 months to <2 years of age.

All patients in each cohort will be administered a single dose of dalbavancin in addition to background anti infective treatment to be chosen by the investigator according to standard of care. Pharmacokinetic samples will be obtained at various timepoints. Dalbavancin can be administered at any time (before, during or after) the standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients who will be receiving at least 24 hours of appropriate non-investigational intravenous anti-infective treatment for known or suspected bacterial infections with the exception of urinary tract infections.
* Written parental informed consent.
* Able to comply with the protocol for the duration of the study.
* Expected to survive throughout the study.
* Normal audiologic assessment within 3 days prior to the study drug infusion.

Exclusion Criteria:

* Investigational drug within 30 days or 5 half-lives, whichever is longest, preceding the first dose of study medication.
* History of fluctuant hearing, persistent tinnitus, balance disorder, otologic surgery or disease, tumor of the head, neck, or auditory system, head injury, Meniere's disease, autoimmune inner ear disease, perilymphatic fistula, CNS disorder resulting in hearing deficits, or significant noise exposure.
* Significant exposure to aminoglycoside antibiotics or chemotherapy currently or within a week prior to enrollment into the study or current use of loop diuretics.
* Patients continuing on vancomycin treatment or are anticipated to begin vancomycin or other glycopeptide treatment during the 7 day period after dalbavancin administration.
* Patients with any clinically significant abnormality other than that associated with their underlying disease. Aminotransferases (AST, ALT) >5 x ULN; total bilirubin and alkaline phosphatase) >2 x ULN.
* Albumin < half lower limit of normal or physical exam evidence of malnutrition.
* Patients who are less than one year of age, and were born with gestational age of less than 32 weeks.
* Positive urine (or serum) pregnancy test at screening (post menarchal females only) or after admission (prior to dosing).
* Known to have hypersensitivity to glycopeptides.
* Calculated creatinine clearance <30 ml/min using the Schwartz method.
* Pregnant or nursing females.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Ages: 3 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics in pediatric patients by measuring AUC 0-inf of dalbavancin. | At 0.5 hours, 4 hours, 12 hours, 24 hours,144 hours and 648 hours post-dose.
  To characterize the pharmacokinetics of dalbavancin in pediatric patients aged 3 months to 11 years (inclusive) following the intravenous administration of a single dose of dalbavancin.
To characterize the pharmacokinetics in pediatric patients by measuring Cmax of dalbavancin. | At 0.5 hours, 4 hours, 12 hours, 24 hours,144 hours and 648 hours post-dose.
  To characterize the pharmacokinetics of dalbavancin in pediatric patients aged 3 months to 11 years (inclusive) following the intravenous administration of a single dose of dalbavancin.
To characterize the pharmacokinetics in pediatric patients by measuring AUC0-last of dalbavancin. | At 0.5 hours, 4 hours, 12 hours, 24 hours,144 hours and 648 hours post-dose.
  To characterize the pharmacokinetics of dalbavancin in pediatric patients aged 3 months to 11 years (inclusive) following the intravenous administration of a single dose of dalbavancin.
To characterize the pharmacokinetics in pediatric patients by measuring AUC0-t of dalbavancin. | At 0.5 hours, 4 hours, 12 hours, 24 hours,144 hours and 648 hours post-dose.
  To characterize the pharmacokinetics of dalbavancin in pediatric patients aged 3 months to 11 years (inclusive) following the intravenous administration of a single dose of dalbavancin.
To characterize the pharmacokinetics in pediatric patients by measuring Tmax of dalbavancin. | At 0.5 hours, 4 hours, 12 hours, 24 hours,144 hours and 648 hours post-dose.
  To characterize the pharmacokinetics of dalbavancin in pediatric patients aged 3 months to 11 years (inclusive) following the intravenous administration of a single dose of dalbavancin.
To characterize the pharmacokinetics in pediatric patients by measuring t1/2 of dalbavancin. | At 0.5 hours, 4 hours, 12 hours, 24 hours,144 hours and 648 hours post-dose.
  To characterize the pharmacokinetics of dalbavancin in pediatric patients aged 3 months to 11 years (inclusive) following the intravenous administration of a single dose of dalbavancin.

SECONDARY OUTCOMES:
To evaluate the safety of a single dose of dalbavancin which will be measured by adverse event monitoring. | one year
To evaluate the safety of a single dose of dalbavancin which will be measured by clinical laboratories (hematology and serum chemistry). | one year
To evaluate the safety of a single dose of dalbavancin which will be measured by blood pressure and pulse rate. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunne, MD, Study Director — Durata Therapeutics
Locations (12):
- United States (10):
  - University Arkansas Medical Center, Little Rock, Arkansas
  - University of California, San Diego, San Diego, California
  - Connecicut Children's Hospital, Hartford, Connecticut
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Columbia University, New York, New York
  - Duke Medical Center, Durham, North Carolina
  - Pediatric Pharmacology, Toledo, Ohio
  - Texas Children's Hospital - Clinical Care Center, Houston, Texas
- Estonia (2):
  - Tallin's Children Hospital Pediatric Clinic, Tallinn
  - Tartu University Hospital Anesthesiology & Intensive Care, Tartu